CLINICAL TRIAL: NCT02069054
Title: Relationship Between Airway Inflammation and Remodeling in Asthma and COPD Patients.
Brief Title: Airway Inflammation and Remodeling in Asthma and COPD.
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: IPU-DIMPA-WUM13(2)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2014-02

CONDITIONS: Asthma; COPD
Keywords: asthma; COPD; airway inflammation; remodeling; cytokines; airway wall thickness
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — induced sputum, BALF, bronchial mucosa samples, exhaled breath condensate, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: Patients with mild to moderate asthma diagnosed in accordance with GINA
- COPD: Patients with mild to moderate COPD diagnosed in accordance with GOLD
- Control: Healthy subjects

SUMMARY:
Asthma and chronic obstructive pulmonary disease (COPD) are inflammatory airway diseases. Although the clinical features of asthma and COPD may be similar, the pathogenesis of these diseases differs in many aspects.

The aim of this study is:

* to evaluate airway inflammation in asthma and COPD,
* to evaluate airway remodeling in asthma and COPD as compared to healthy subjects,
* to assess the relationship between markers of airway inflammation and airway remodeling in asthma and COPD patients.

Material and methods:

* mild to moderate asthma patients diagnosed in accordance with Global Initiative for Asthma (GINA) guidelines,
* mild to moderate COPD patients diagnosed in accordance with Global initiative for chronic Obstructive Lung Disease (GOLD) guidelines,
* healthy subjects as controls.

Airway inflammation is assessed in induced sputum (IS), exhaled breath condensate (EBC), bronchoalveolar lavage fluid (BALF) and specimens from endobronchial forceps biopsy. Airway wall thickness is evaluated in high resolution computed tomography (HRCT), endobronchial ultrasound (EBUS) and basement membrane thickness (BMT) in biopsy specimens.

We plan to compare airway inflammation and features of airway remodeling in asthma and COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of asthma or COPD in accordance with GINA or GOLD, respectively
* control group - healthy volunteers without any history of lung disease

Exclusion Criteria:

* age below 18 years
* exacerbation in the past 6 weeks
* inhaled corticosteroid therapy at least 6 weeks prior to study enrollment
* significant co-morbidities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with stable asthma and COPD invited to Clinical Hospital in Warsaw
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Approximately 1-2 months after completion of study procedures (bronchoscopy, induced sputum, etc.) in all patients (probably January 2015)
  Inflammatory markers in exhaled breath condensate and induced sputum in healthy subjects, COPD and asthma patients.
Airway wall thickness | Approximately 1-2 months after completion of study procedures (bronchoscopy with EBUS, HRCT) in all patients (probably January 2015)
  Airway wall thickness in healthy subject, COPD and asthma patients assessed by HRCT and EBUS

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergology, Medical University of Warsaw 02-097, Warsaw, Poland